CLINICAL TRIAL: NCT04336124
Title: A Phase I Safety and Pharmacokinetic Study of CVM-1118 Extended-Release Capsules Administered Orally to Patients With Advanced Cancers
Brief Title: Safety and Pharmacokinetic Study of CVM-1118 Extended-Release in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVMEX-001
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Advanced Cancer
Keywords: Oncology; Advanced Solid Malignancy; Tumor Response; Safety and pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — Capsules

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVM-1118 ER (Experimental): Dose escalation (escalation from 400, 600, 800 to 1200 mg of CVM-1118 ER Capsule)
  Interventions: Drug: CVM-1118 Extended-Release (ER) Capsules (200 mg/capsule)

INTERVENTIONS:
Drug: CVM-1118 Extended-Release (ER) Capsules (200 mg/capsule) — Patients will receive initial dose regimen: 400 mg of CVM-1118 ER Capsule per day (200 mg BID) in a 28-day cycle for 4 cycles.
  Dose escalates from 400, 600, 800, to 1200 mg of CVM-1118 ER capsules with either BID or TID dosing.
  A single-patient cohort per dose level (accelerated titration design) will be applied to the first two cohorts, 400 and 600 mg daily, and followed by the conventional 3+3 dose escalation design from the dose level of 800 mg/day.
  If 2 or more patients experience a DLT, no further dose escalation will occur.
  Other Names: TRX-818 ER

SUMMARY:
CVM-1118 Immediate-release (IR) Capsule and CVM-1118 Extended-release (ER) Capsule are proprietary oncology products developed by TaiRx, Inc. for the treatment of patients suffering from advanced cancer. Due to the short elimination half-life of CVM-1118 IR capsules, the extended release (ER) formulation, containing mini-tablets in hard capsule, has been developed to prolong the drug absorption and longer exposure after oral administration. The designed dose of CVM-1118 ER was 200 mg per capsule to provide a more patient-compliant and safe dosage of CVM-1118. The clinical study CVMEX-001 is therefore designed to evaluate the safety and pharmacokinetics of CVM-1118 extend release (ER) Capsule (200 mg/capsule) in patients with advanced cancer.

DETAILED DESCRIPTION:
The CVM-1118 ER Capsule will be orally administered BID or TID before meal in 28-day treatment cycles. Patients will receive 400, 600, 800 to 1,200 mg of CVM-1118 ER Capsule in sequential cohort based on safety and dose tolerability. A single-patient cohort per dose level (accelerated titration design) will be applied to the first two cohorts, 400 and 600 mg daily, and followed by the conventional 3+3 dose escalation design from the dose level of 800 mg/day. Within the first two cohorts, if any Grade 2 or greater toxicity at least possibly attributable to CVM-1118 ER capsule is reported in the first patient during first cycle, a single-patient cohort will be converted to conventional 3+3 study design once and expand to a minimum of 3 evaluable patients for assessment of toxicity within the first cycle. Dose escalation will occur until DLT occurs in 2 or more patients within a dose level. In any cohort, if 1 patient experiences a DLT, 3 additional patients will be enrolled to that dose level. If 2 or more patients experience a DLT, no further dose escalation will occur. Plasma pharmacokinetics samples will be collected at pre-determined time-points for all patients participating in the dose-escalation study.

This study will be completed and closed once the MTD is determined for CVM-1118 ER capsules. However, at the end of 4 cycles, it is recommended that some patients should continue receiving the clinical benefit from CVM-1118 ER capsules. Thus, patients may be continuously treated at the assigned dose level or next higher dose level provided it has been shown to be safe in a previously treated cohort by safety committee, until the treating physician feels the patient is no longer benefiting from the treatment, or CVM-1118 ER Capsule becomes commercially available, as applicable in the country in which the patient lives. In the event of unacceptable toxicity at a given dose, CVM-1118 can be reduced to the previous dose level or suggested lower dose by PI. If unacceptable toxicity persists despite 2 dose reductions, the patient should be removed from study.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor eligibility:

   Histologically or cytologically confirmed advanced malignancies, which is refractory to standard of care therapy, or for whom no standard of care therapy is available.
2. Solid tumors must have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy. Lymphomas must have measurable disease as per Revised Response Criteria for Malignant Lymphomas.
3. ECOG performance status 0 to 2. Resolution of all acute toxic effects of prior therapy or surgical procedures to grade 1 (except alopecia).
4. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
   2. Total serum bilirubin ≤1.5 x ULN (except for patients with documented Gilbert's syndrome)
   3. Absolute neutrophil count (ANC) 1,500/µL
   4. Platelets 90,000/µL
   5. Hemoglobin 9.0 g/dL
   6. Serum creatinine ≤1.5 x ULN or creatinine clearance of ≥ 60 mL/min
5. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the study prior to enrollment.
6. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients presenting with any of the following will not be included in the study:

   1. Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of starting study treatment.
   2. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue except for patients with lymphoma
   3. Current treatment on another clinical study.
   4. Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
2. Any of the following within 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and sponsor, the 6-month post-event-free period for a patient with a pulmonary embolus can be waived if due to advanced cancers. Appropriate treatment with anticoagulants is permitted.
3. Hypertension that cannot be controlled by medications (>160/100 mmHg despite optimal medical therapy).
4. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily is allowed).
5. Known human immunodeficiency virus infection.
6. Hepatitis B virus (HBV) or hepatitis C virus (HCV) with evidence of chronic active disease or receiving/requiring antiviral therapy.
7. History of receiving organ transplantation or immune disorders that require continuous immunosuppressant agent therapy.
8. Pregnancy or breastfeeding. Female patients must be surgically sterile or be post-menopausal or must agree to the use of effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
9. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the patient inappropriate for entry into this study.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of CVM-1118 ER Capsule | up to 28 days
  Dose escalation will occur until DLT occurs in 2 or more patients within a dose level. In any cohort, if 1 patient experiences a DLT, 3 additional patients will be enrolled to that dose level. If 2 or more patients experience a DLT, no further dose escalation will occur.
Maximum tolerated dose (MTD) of CVM-1118 ER Capsule | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a DLT after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT. The Safety Committee may expand the cohort beyond six patients to better define the safety profile of this cohort in the search for the MTD.

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity of CVM-1118 ER Capsule | up to 56 days
  RECIST 1.1 for solid tumor and Revised Response Criteria for Malignant Lymphoma
Measure of plasma pharmacokinetic (PK) profiles of CVM-1118 and its metabolite CVM-1125 to include AUC(0-last) | Cycle 1 Day 1 and Day 15: pre-dose, 2, 3.5, 5, 7, 9, and 12 hours post dose
  AUC(0-last): area under the plasma concentration versus time curve to the time of the last measurable concentration
Measure of plasma pharmacokinetic (PK) profiles of CVM-1118 and its metabolite CVM-1125 to include Cmax | Cycle 1 Day 1 and Day 15: pre-dose, 2, 3.5, 5, 7, 9, and 12 hours post dose
  Cmax: Maximum plasma concentration
Measure of plasma pharmacokinetic (PK) profiles of CVM-1118 and its metabolite CVM-1125 to include Tmax | Cycle 1 Day 1 and Day 15: pre-dose, 2, 3.5, 5, 7, 9, and 12 hours post dose
  Tmax: Time to maximum plasma concentration
Measure of plasma pharmacokinetic (PK) profiles of CVM-1118 and its metabolite CVM-1125 to include T(1/2) | Cycle 1 Day 1 and Day 15: pre-dose, 2, 3.5, 5, 7, 9, and 12 hours post dose
  T(1/2): Terminal elimination half-life
Time to tumor progression (TTP) | up to 112 days
  Time to progression (TTP) is defined as the time from the first dose of study drug to the time of progression

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, M.D., Principal Investigator — National Cheng Kung University Hospital,Taiwan; Li-Yuan Bai, M.D., Principal Investigator — China Medical University Hospital
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan